CLINICAL TRIAL: NCT05739812
Title: The Efficacy and Safety of Chinese Domestic Surgical Robot System in Urological Telesurgery, an Exploratory Study
Brief Title: The Efficacy and Safety of Chinese Domestic Surgical Robot System in Urological Telesurgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Haitao Niu, MD, Professor Haitao Niu (the department of Urology), The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SDWG-NST600S-YCSS-5
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Renal Cell Carcinoma; Adrenal Tumor; Nonfunctioning Kidney; Renal Pelvis Carcinoma; Ureteral Tumor; Bladder Cancer; Prostate Cancer; Pelvic Tumor; Renal Cyst; Duplex Kidney; Renal Calculi; Ureteral Calculi; Ureteropelvic Junction Obstruction; Penile Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Adrenal Gland Neoplasms; Ureteral Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Pelvic Neoplasms; Kidney Calculi; Ureteral Calculi; Multicystic renal dysplasia, bilateral; Penile Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urological disease group (Experimental): Patients with urological diseases (renal cell carcinoma, nonfunctioning kidney and adrenal tumor, renal pelvis carcinoma, ureteral tumor, bladder cancer, prostate cancer, pelvic tumor) will be treated by telesurgery.
  Interventions: Device: telesurgery by domestic surgical robot

INTERVENTIONS:
Device: telesurgery by domestic surgical robot — telesurgery of urological diseases by domestic surgical robot

SUMMARY:
A single-arm clinical trial was designed in this study. The surgeon will perform urological telesurgery for patients using Chinese domestically produced "MicroHand S" surgical robot system. The "MicroHand S" surgical robot system consists of two physically separated subsystems named the "surgeon console" and the "patient side cart". The surgeon console includes a stereo image viewer, two master manipulators, a control panel and several foot pedals. The patient side cart includes a passive arm that can slide in the up-down direction and be adjusted forward and backward, a swivel head that can rotate around the vertical axis, and three slave arms. In addition, surgical instruments and sterile bags are the essential accessories for the "patient side cart". The principle of the telesurgery is as follows: the surgeon console takes the surgeon's input and translates manipulation into a control signal. After network transmission, the signals will be received by the patient side cart and will be used to control the slave robot to manipulate the instruments to perform the operation within the patient's cavity. The 3D images captured by the endoscopic camera will be simultaneously sent back to the screen of the surgeon console as visual feedback. Data between the surgeon console and the patient side cart will be transmitted through a 5G network or other advanced network networking scheme. The surgeon remotely manipulates the slave arms and performs surgeries for patients in remote areas. The safety and efficacy of the robot system in remote clinical treatment will be verified by the primary and the secondary evaluation criteria. One hundred patients with urological diseases will be enrolled in the clinical trial.

Primary evaluation criterion:

The success rate of the surgery. Surgery success is defined as that all surgeries are performed remotely and safely without transfering to other types of surgery, such as open surgery or normal robot-assisted surgery.

Secondary evaluation criteria:

Operative time, blood loss, postoperative pain, preoperative adjusting time, hospitalization time, average network latency, task load, peer recognition, anxiety index.

Patient enrollment:

This experiment aims to investigate the safety and effectiveness of the domestic robot system in clinical urological surgery under the current network networking scheme. It is planned that 100 patients with urinary system diseases will participate in the clinical trial.

DETAILED DESCRIPTION:
Objective: This clinical trial aims to evaluate the efficacy and safety of telesurgery for patients with urological tumors using Chinese independently developed "MicroHand S" Surgical Robot System under the current advanced network networking scheme.

Content: A single-arm clinical trial was designed in this study. The product is domestically produced "MicroHand S" surgical robot system (Shandong Weigao Surgical Robot Co., Ltd, China). The patients will be fully informed and the written informed consent will be signed before the clinical study, According to the inclusion criteria and exclusion criteria, the researchers will conduct a detailed screening to determine whether the patients are suitable for the clinical study. Telesurgery will be conducted for patients who meet the inclusion criteria using the "MicroHand S" surgical robot system. Data between the "surgeon console" and the "patient side cart" will be transmitted through the current advanced network networking scheme. Fifty telesurgeries has been performed for patients with renal tumor, adrenal tumor, or nonfunctional kidney disease in 2021. All the surgeries were completed successfully, which made an positive social influence. In order to explore other indications, 100 subjects will be enrolled in the clinical trial. All diseases will be included if it is applicable to be treated by telesurgery, such as, adrenal tumor, renal tumor, renal cyst, duplex kidney, renal calculi, ureteral calculi, ureteropelvic junction obstruction (UPJO), nonfunctional kidney, renal pelvis tumor, ureteral tumor, bladder cancer, prostate cancer, pelvic tumor, penile cancer, etc. The safety and efficacy of remote clinical treatment using the domestic robot system will be verified according to the primary evaluation criterion, secondary evaluation criteria, and safety evaluation index.

Network connection plan: Two network connection plans were designed in advance to transmit data between the two sites (the master and the slave) in telesurgery. Plan A: Both signals (the control signals and the video signals) were transmitted in a VPN encryption mode under 5G wireless network or other advanced network networking scheme. Plan B: Both signals were transmitted through the dedicated line. When 5G network or other advanced network networking scheme was unstable and the surgery was affected, Plan A could be switched to Plan B to ensure the success of telesurgery. The two sites were also connected through a video conference system for real time communication and coordination.

Primary evaluation criterion: The primary evaluation criterion is the success rate of the surgery.

Secondary evaluation criteria: Secondary evaluation criteria include operative time, intraoperative blood loss, assembly time, postoperative pain, hospital stay, time to first flatus, average network latency, task load index, patient acceptance of telesurgery, peer surgeon acceptance of telesurgery, patient anxiety index, surgeon anxiety index.

Safety evaluation index: (1) Organ and vascular injury events related to the robot, including the following injury events: a. Whether there is adjacent organ injury caused by the robot functional failure during the operation, including liver, spleen and intestinal injury; b. Whether there is hemorrhoea caused by vascular injury caused by the robot functional failure during the operation. (2) Adverse events during the study. (3) Instrument malfunction. a. The communication between the "surgeon console" and the "patient side cart" is strongly disturbed, the slave arms fail to move and malfunction cannot be eliminated after reset and restart. b. by surgical instruments cannot be loosened after the tissue is clamped. c. An alarm sounds when install the instruments. d. Instruments lose efficacy or they are damaged. (4) Vital signs (body temperature, blood pressure, and heart rate). (5) Laboratory examination: blood routine, liver and kidney function, electrolyte.

Researcher selection: In order to strictly ensure the homogeneity and uniformity of researchers, operators are required to have certain qualifications. All surgeons must have at least 5 years of experience in laparoscopic general surgery and at least 1-year experience in robotic surgery. The surgeon will be trained in delay simulation training before the trial. Meanwhile, product training is also required before the trial, and each surgeon must complete at least 20 surgeries with the tested robot. All the trainings above are to help surgeons cross the learning curve.

Background: With the combination of robotic and network communication technology, telesurgery has become a reality. On the one hand, telesurgery can conserve and optimize medical resources, providing high-quality medical services to unbalanced areas, such as rural areas, stricken areas and battlefields. On the other hand, telesurgery can reduce the time spent by patients waiting for treatment and thus prevent diseases from worsening. In recent years, the rapid advancements of the fifth and sixth generation network communication technologies and surgical robotic devices have again boosted the development of telesurgery since the Lindbergh operation and the research of Anvari et al. Especially in a country as vast as China, where the difference of the level of medical care between developed cities and rural areas is huge and the need for telesurgery is enormous. The demand for telemedicine has also risen significantly, particularly since the outbreak of COVID-19. However, as the most challenging components of telemedicine, telesurgery has still developed slowly, and most studies of it are limited to single-center experiences and as such have some inherent limitations. Based on this background, we have successfully conducted preliminary studies in which we verified the safety and feasibility of multiple network plans for telesurgery such as 5G network slicing technology and heterogeneous multilink network converged transmission technology.

In 2021, our research group carried out a multicenter prospective study evaluating efficacy and safety of telesurgery for upper urological tumors using the "Micro Hand S" system robot and a 5G network in Shandong Province, China.

With the prevalence of telesurgery, indications should not limited in upper urological diseases. More indications should be explored. On such basis, this clinical trial was designed and performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years.
* BMI was 18-30 kg/m2.
* The American Society of Anesthesiologists (ASA) classification was I, II, or III.
* Patients with adrenal tumor that need radical or partial adrenalectomy (nonfunctioning adenoma, < 5cm in diameter).
* Patients with renal cell carcinoma that need radical nephrectomy or partial nephrectomy.
* Patients with renal cyst that need decompression surgery.
* Patients with duplex kidney that need radical nephroureterectomy.
* Patients with renal calculi that need intrasinusal pyelolithotomy.
* Patients with ureteral calculi that need ureterolithotomy.
* Patients with ureteropelvic junction obstruction (UPJO) that need pyeloplasty.
* Patients with urological diseases (such as, pelvic segment disease of the ureter, or duplex kidney) that need ureteral reimplantation.
* Patients with nonfunctioning kidney that need radical nephrectomy.
* Patients with renal pelvis carcinoma that need radical nephroureterectomy.
* Patients with ureteral tumor that need radical nephroureterectomy.
* Patients with bladder cancer that need radical or partial cystectomy.
* Patients with prostate cancer that need radical prostectomy.
* Patients with penile cancer that need Ilioinguinal lymph node dissection.

Exclusion Criteria:

* Women in pregnancy or lactation
* A history of epilepsy or mental illness
* Previous relevant operation history (all abdominal operations that may increase difficulty in telesurgery)
* Patients with a severe cardiovascular and cerebrovascular disease with New York Heart Association (NYHA) classification III-IV and pulmonary insufficiency who cannot tolerate the operation
* Liver cirrhosis, kidney failure and other severe liver and kidney dysfunction (ALT and AST exceeded 3 times of the upper limit of normal value, Cr exceeded 1.5 times of the upper limit of normal value)
* Patients with general hemorrhagic diseases and coagulation dysfunction (prothrombin activity, PTA <25%)
* Patients with active hepatitis and AIDS
* Patients with uncorrected diabetes (random blood glucose, RBG >11.1 mmol/L) and hypertension (≥160/100 mmHg)
* Patients with severe allergic constitution and suspected or confirmed alcohol, medicine or drug addiction
* Patients with abdominal infection, peritonitis or diaphragmatic hernia
* Patients with severe systemic infection or metastatic disease
* Patients who are unable to voluntarily participate and sign informed consent
* Other circumstances under which the investigator considers it is inappropriate to participate in this clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
success rate of the telesurgery | after the study is completed, up to 2 years.
  The success of the telesurgery is the robot-assisted telesurgery without transfering to other types of surgery, such as open surgery or normal robot-assisted surgery. The number of the success divided by the total number is the success rate.

SECONDARY OUTCOMES:
Operative time | after each procedure is completed, all data will be collected within 4 months
  The operative time is from the time the robot is assembled till the incision is sutured.
Intraoperative blood loss | after each procedure is completed, all data will be collected within 4 months
  Intraoperative blood loss is the total amount of blood loss from the beginning of the operation (after the robot is assembled) to the incision is sutured. The blood loss is estimated by weight. Estimated blood loss (g) = the weight of the gauze wiping up all the blood - the weight of the dry gauze. And 1g = 1ml.
Postoperative pain | at 24±2 hours after each procedure is completed, all data will be collected within 4 months
  Postoperative pain is assessed by a visual analog scale (VAS) with a range from 0 point (no pain) to 10 points (maximum pain) at 24±2 hours postoperatively.
Assembly time | from the time the robot starts to the time the trocar is connected to the robot arm during each procedure, all data will be collected within 4 months
  The assembly time is from the time the robot starts to the time the trocar is connected to the robot arm.
Hospital stay | from admission to discharge for each patients, all data will be collected within 4 months
  The hospital stay is the total number of days from the admission to the discharge of patients.
Average network latency | during the whole procedure in each telesurgery, all data will be collected within 1 months
  Average network latency is monitored by specific software in real time during the telesurgery.
Task load | after each procedure is completed, all data will be collected within 4 months
  Task load will be evaluated through NASA-TLX questionnaire filled by the surgeons.
Patient acceptance | one day before the telesurgery, all data will be collected within 4 months
  Patient acceptance of telesurgery will be assessed through TPSQ questionnaire filled by the patients 1 day before operation.
Peer surgeon acceptance | one day before the telesurgery, all data will be collected within 4 months
  Peer surgeon acceptance of telesurgery will be systematic reviewed through TAKA questionnaire filled by peer surgeons.
Patient anxiety index | one day before or after the telesurgery, all data will be collected within 4 months
  Patient anxiety index will be assessed through TP-SAS questionnaire filled by patients.
Surgeon anxiety index | one day before or after the telesurgery, all data will be collected within 4 months
  Surgeon anxiety index will be assessed through TP-SAS questionnaire filled by operating surgeons and assistant surgeons.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Niu, PhD, Study Chair — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen H, Pan X, Yang J, Fan J, Qin M, Sun H, Liu J, Li N, Ting DSW, Chen Y. Application of 5G Technology to Conduct Real-Time Teleretinal Laser Photocoagulation for the Treatment of Diabetic Retinopathy. JAMA Ophthalmol. 2021 Sep 1;139(9):975-982. doi: 10.1001/jamaophthalmol.2021.2312. PMID 34236391
- [Background] Tian W, Fan M, Zeng C, Liu Y, He D, Zhang Q. Telerobotic Spinal Surgery Based on 5G Network: The First 12 Cases. Neurospine. 2020 Mar;17(1):114-120. doi: 10.14245/ns.1938454.227. Epub 2020 Mar 31. PMID 32252160
- [Background] Nguan C, Miller B, Patel R, Luke PP, Schlachta CM. Pre-clinical remote telesurgery trial of a da Vinci telesurgery prototype. Int J Med Robot. 2008 Dec;4(4):304-9. doi: 10.1002/rcs.210. PMID 18803341
- [Background] Sterbis JR, Hanly EJ, Herman BC, Marohn MR, Broderick TJ, Shih SP, Harnett B, Doarn C, Schenkman NS. Transcontinental telesurgical nephrectomy using the da Vinci robot in a porcine model. Urology. 2008 May;71(5):971-3. doi: 10.1016/j.urology.2007.11.027. Epub 2008 Mar 4. PMID 18295861
- [Background] Marescaux J, Leroy J, Rubino F, Smith M, Vix M, Simone M, Mutter D. Transcontinental robot-assisted remote telesurgery: feasibility and potential applications. Ann Surg. 2002 Apr;235(4):487-92. doi: 10.1097/00000658-200204000-00005. PMID 11923603
- [Background] Yi B, Wang G, Li J, Jiang J, Son Z, Su H, Zhu S, Wang S. Domestically produced Chinese minimally invasive surgical robot system "Micro Hand S" is applied to clinical surgery preliminarily in China. Surg Endosc. 2017 Jan;31(1):487-493. doi: 10.1007/s00464-016-4945-3. Epub 2016 May 18. PMID 27194259
- [Background] Yao Y, Liu Y, Li Z, Yi B, Wang G, Zhu S. Chinese surgical robot micro hand S: A consecutive case series in general surgery. Int J Surg. 2020 Mar;75:55-59. doi: 10.1016/j.ijsu.2020.01.013. Epub 2020 Jan 23. PMID 31982634